CLINICAL TRIAL: NCT03869164
Title: Multi-center Trial of Transcatheter Edge-to-edge Mitral Valve Repair With ValveClamp System in High Risk Patients With Degerative Mitral Regurgitation
Brief Title: Multi-center Trial of ValveClamp
Acronym: CLAMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YL-2018-27
Record Dates: First submitted 2019-02-25; First posted 2019-03-11 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Evaluate the Safety and Efficacy of the ValveClamp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ValmpClamp Arm (Experimental)
  Interventions: Device: ValveClamp

INTERVENTIONS:
Device: ValveClamp — ValveClamp is an easy-to-operate transcatheter edge-to-edge mitral valve repair system with larger coaptation width

SUMMARY:
The ValveClamp (Hanyu Medical Technology, Shanghai, China) is the first edge-to-edge mitral valve repair system for interventional operation in China, which is composed of the front clamp, the rear clamp and the closed ring. The purpose of the multi-center trial is to evaluate the safety and efficacy of the ValveClamp for degenerative mirtal regurgistation.

DETAILED DESCRIPTION:
The transcatheter edge-to-edge mitral valve repair device MitraClip (Abbott Vascular, Santa Clara, CA, USA) is the most mature device for mitral regurgitation. Another transcatheter edge-to-edge mitral valve repair device, the PASCAL system, has been shown to be feasible to reduce MR severity. Both the MitraClip and PASCAL devices need a complex steerable deliver system and thus complex process to steer the device to mitral valve. An easy-to-operate transcatheter edge-to-edge mitral valve repair system (ValveClamp) with larger coaptation width was thus recently developed in China. The ValveClamp (Hanyu Medical Technology, Shanghai, China) is the first edge-to-edge mitral valve repair system for interventional operation in China, which is composed of the front clamp, the rear clamp and the closed ring. The purpose of the multi-center trial is to evaluate the safety and efficacy of the ValveClamp for degenerative mirtal regurgistation.

ELIGIBILITY:
Inclusion Criteria:

1. age older than 60 years;
2. moderate to severe or severe mitral regurgitation;
3. symptoms (New York Heart Association [NYHA] cardiac function class ≥2) related to MR;
4. the primary regurgitant jet originated from malcoaptation of the A2 and P2 scallops of the mitral valve;
5. high risk for surgery according the MVARC criteria;
6. providing signed informed consent.

Exclusion Criteria:

1. acute myocardial infarction in the prior 4 weeks of the intended treatment;
2. any interventional or surgical cardiac procedure performed within 30 days prior;
3. the need for any other cardiac surgery;
4. echocardiographic evidence of intracardiac mass, thrombus, or vegetation;
5. life expectancy within 12 months;
6. moderate or severe aortic stenosis or regurgitation;
7. mitral valve orifice area <3.5 cm2;
8. untreated significant coronary stenosis;
9. history of mitral valvuloplasty;
10. Infective endocarditis and rheumatic heart disease;
11. untreated cardiogenic shock, acute pulmonary congestion;
12. unfavored mitral valve anatomy that may preclude device implantation including: calcification or significant cleft in area of the A2 and/or P2 scallops, significant regurgitation beyond A2 or P2 scallops and short posterior leaflet (<10mm).
13. Other clinical trials that the subjects participated in have not reached the end point.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2021-12-13 (Estimated); Study Completion 2025-12-08 (Estimated)

PRIMARY OUTCOMES:
The device success rate | 12months
  freedom from the composite end point of death from any cause, surgery for valve dysfunction, and MR ≥3+ at one month.

SECONDARY OUTCOMES:
Incidence of adverse cardiovascular events | immediate post-operation
  death, severe arrhythmia, pericardial tamponade, emergency surgery, cardiac shock, endocarditis, bleeding , and other complications caused by procedure
Incidence of deaths | 1,6,12months
  All cause deaths (cardiac death, and non cardiac death) or strokes
Incidence of mitral valve re-surgery | 1,6,12months
  Mitral valve re-surgery because of the failure of operation, embolism, clamp's falling off.
Grading of mitral regurgitation by echocardiography | 1,6,12months
  The echocardiographic analysis was performed according to the American Society of Echocardiography guidelines. The severity of MR was graded as none or trac e (0+), mild(1+), moderate(2+), moderate to severe (3+) or severe (4+) by using the EVERST criteria.
New York Heart Association (NYHA) class | 1,6,12months
  The NYHA cardiac function class containing the levels of Ⅰ, Ⅱ, Ⅲ, Ⅳ, relies on the concept of ordinary physical activities. Class Ⅰ means that patients have cardiac disease but without the resulting limitations of physical activity. Class Ⅱ means that patients have cardiac disease resulting in slight limitation of physical activity. Class Ⅲ refers to that patients have cardiac disease resulting in marked limitation of physical activity. Class Ⅳ refers to that patients have cardiac disease resulting in inability to carry on any physical activity without discomfort.
brain natriuretic peptide | 1,6,12months
  BNP is a kind of laboratory blood test index to reflect the cardiac function.
severe adverse events | 1,6,12months
  Severe adverse events include injury of mitral valves, re-inpatient for poor cardiac function and other severe adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Wenzhi Pan, M.D., Principal Investigator — Department of Cardiology, Zhongshan Hospital, Fudan University
Locations (1):
- Zhongshan Hopital of Fudan University, Shanghai, Shanghai, China, China